CLINICAL TRIAL: NCT00688207
Title: An Open Label Single Oral Dose Study in Patients With Mild Alzheimer's Disease to Assess the Pharmacokinetics of Extended Release Formulation of Rosiglitazone (RSG XR) in This Population
Brief Title: Mild Alzheimer''s Disease to Assess the of Extended Release Formulation of Rosiglitazone (RSG XR)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA109941
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Alzheimer's Disease
Keywords: PPAR agonist,; Rosiglitazone XR,; BRL-049653.; Alzheimer's disease,
MeSH Terms: conditions — Alzheimer Disease | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosiglitazone (Experimental): An open-label, single, oral dose of 4mg of rosiglitazone in the morning under fasted conditions
  Interventions: Drug: Rosiglitazone (Extended Release)

INTERVENTIONS:
Drug: Rosiglitazone (Extended Release) — open-label, single, oral, 4mg dose

SUMMARY:
The present pharmacokinetic study is designed to assess the pharmacokinetics of RSG XR as monotherapy in patients with mild Alzheimer's disease (AD) as such information will not be obtained from the current phase III trials . The study aims to enroll fourteen patients (seven of each APOE genotype). Each patient will receive a single oral dose of 4mg of RSG XR in the morning under fasted conditions and PK samples will be taken up to 36h.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a clinical diagnosis of probable Alzheimer's disease in
* accordance with NINCDS-ADRDA3 criteria for at least 3 months
* Subject has mild Alzheimer's disease as defined by a MMSE score 18 to 26 inclusive
* at Screening
* Hachinski Ischemia Score ≤ 4 at Screening
* Subjects aged ≥50 and ≤90 years.
* Subject has not taken an approved Alzheimer's therapy in the last 30 days.
* Current use of medication is in accordance with the criteria listed in Section 9.1).
* Female subjects must be post-menopausal (i.e. >1 year without menstrual period),
* surgically sterile, or agree to use adequate method of contraception for the duration of the study.
* Female subjects who are pre-menopausal or who have been postmenopausal for <1 year must undertake pregnancy testing at screening, which must
* be negative. More than one pregnancy test may be required (i.e., when the time period between enrolment and study treatment is > 7 days).
* Pregnancy testing will be performed at screening, pre-dose (Day 1) and follow-up visit for all women of child-bearing potential and those who have been postmenopausal for less than 1 year. If clinically indicated, a urine or serum pregnancy test may be performed at anytime during the study.
* Brain CT or MRI scan performed within the past 12 months or at Screening, showing no evidence of any other potential cause of dementia other than Alzheimer's disease.
* Neurological exam without focal changes (excluding changes attributable to AD or peripheral trauma).
* Subjects who live with or who have a regular caregiver who is willing to attend all visits, oversee the subject's compliance with the protocol specified procedures and study medication, and who is willing to report on subject's status.
* Subject has provided full written informed consent prior to the performance of any protocol-specified procedure.
* Subjects considered for enrolment must have a QTc (either QTc B (Bazett's
* correction) or QTc F (Fridericia's correction)) <450msec at the Screening Visit, with the exception of subjects with bundle branch block (for whom either QTc B or QTc F must be <480msec).

Exclusion Criteria:

* Diagnosis of possible, probable, or definite vascular dementia in accordance with NINDS-AIREN6 criteria
* History or evidence of any other CNS disorder that could be interpreted as a cause of dementia: e.g. cerebrovascular disease (stroke, hemorrhage), structural abnormality, epilepsy, infectious or inflammatory/demyelinating CNS conditions, Parkinson's disease.
* Evidence of the following disorders: current vitamin B12 deficiency, positive syphilis serology or active thyroid dysfunction (particularly that suggestive of hypothyroidism), including abnormally high or low serum levels of thyroid stimulating hormone (TSH) that is clinically significant in the opinion of the investigator.
* History of Type 1 diabetes mellitus or secondary diabetes mellitus.
* Type 2 diabetes mellitus where the subject is being treated with insulin, a PPARγ agonist, or an insulin secretagogue (e.g. a sulfonylurea or glitinide).
* Any patient with an HbA1c ≥8.5%
* History or clinical/laboratory evidence congestive heart failure defined by the New York Heart Association criteria (Class I to IV cardiac status) (Appendix 4).
* History of cardiovascular event within the last 6 months (i.e. intervention, percutaneous coronary intervention, vascular surgery, acute coronary syndrome [non Q-wave myocardial infarction, Q-wave myocardial infarction, unstable angina] or significant arrhythmia; or major intervention (e.g. cardiac surgery or angiography plus stenting) scheduled).
* History of significant psychiatric illness such as schizophrenia or bipolar affective disorder that in the opinion of the Investigator would interfere with participation in the study, major depressive disorder (according to DSM-IV) in the past year, or current active depression requiring initiation of treatment.
* History or presence of gastro-intestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, or any other clinically relevant abnormality, which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* Clinically significant peripheral oedema at the time of screening.
* Current or recent drug or alcohol abuse or dependence (defined by DSM-IV criteria for substance-related disorders), or recent or remote history of the same if that could be a contributing factor to the dementia.
* Systolic blood pressure >165 or <90 mmHg or diastolic blood pressure >95 or <60 mmHg at the time of screening.
* Clinically significant anaemia (i.e. haemoglobin <11 g/dL for males or <10 g/dL for females)
* Patients with GFR ≤50ml/min (assessed by Cockcroft-Gault method ) .
* ALT, AST, or alkaline phosphatase values >2.5 times the upper limit of normal, total bilirubin values >1.5 times the upper limit of normal, or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis, Child-Pugh Class B/C).
* History of a bone marrow transplant.
* Positive hepatitis B virus, hepatitis C virus or HIV test at screening.
* Subject is unable (with assistance, if appropriate) to take study medication or is at risk of non-compliance with study procedures.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
AUC (0-inf) and Cmax of RSG XR | Up to 36 hours

SECONDARY OUTCOMES:
AUC(0-t), t1/2 and tmax for RSG XR | Up to 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: AVA109941 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVA109941 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVA109941 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVA109941 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVA109941 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVA109941 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVA109941 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register